CLINICAL TRIAL: NCT02669264
Title: A Phase 1, Open-label, Adaptive Dose-escalation, Multicenter Study to Evaluate the Tolerability, Safety, Pharmacokinetics, and Anti-tumor Activity of ADCT-402 in Patients With Relapsed or Refractory B-cell Lineage Acute Lymphoblastic Leukemia (B-ALL)
Brief Title: Study of ADCT-402 in Patients With Relapsed or Refractory B-cell Lineage Acute Lymphoblastic Leukemia (B-ALL)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was early terminated prior to part 2 because of slow accrual.
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADCT-402-102
Record Dates: First submitted 2016-01-21; First posted 2016-02-01 (Estimated); Results first posted 2019-09-26 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Loncastuximab tesirine
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — loncastuximab tesirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1: ADCT-402 dose escalation (Experimental): Weekly administration - Participants will receive an intravenous (IV) infusion of ADCT-402, on Days 1, 8, and 15 of each 3-week (21-day) cycle.
  3-week administration - Participants will receive an IV infusion of ADCT-402, on Day 1 of each 3-week (21-day) cycle.
  The dose escalation will be conducted according to a 3+3 design.
  Interventions: Drug: ADCT-402
- Part 2: ADCT-402 expansion (Experimental): All participants will be assigned to the recommended dose and/or schedule of ADCT-402 identified in Part 1 by the Dose Escalation Steering Committee
  Interventions: Drug: ADCT-402

INTERVENTIONS:
Drug: ADCT-402 — Intravenous infusion
  Other Names: Loncastuximab tesirine; Zynlonta

SUMMARY:
This study evaluates ADCT-402 in participants with relapsed or refractory B-cell lineage acute lymphoblastic leukemia (B-ALL). Participants will participate in a dose-escalation phase (Part 1) and dose expansion (Part 2). In Part 2, participants will receive the dose level identified in Part 1.

DETAILED DESCRIPTION:
Study ADCT-402-102 is the first clinical study with ADCT-402 in participants with B-cell lineage acute lymphoblastic leukemia (B-ALL).

ADCT-402 is an antibody drug conjugate (ADC) composed of a humanized antibody directed against human cluster of differentiation 19 (CD19), stochastically conjugated via a valine-alanine cleavable, maleimide linker to a pyrrolobenzodiazepine (PBD) dimer cytotoxin.

The study will be conducted in 2 parts. In Part 1 (dose escalation) participants will receive an infusion of ADCT-402 either on weekly administration or every 3-week administration. participants on weekly administration will receive an infusion of ADCT-402 on Days 1, 8, and 15 of each 3 week treatment cycle. Participants on 3-week administration will receive an infusion of ADCT-402 on Day 1, every 3 weeks. Dose escalation will continue until the maximum tolerated dose (MTD) is determined.

In Part 2 (expansion), all participants will be assigned to the recommended dose and/or schedule of ADCT-402 identified in Part 1 by the Dose Escalation Steering Committee.

For each patient, the study will include a screening period (up to 28 days), a treatment period (until withdrawal), and a follow-up period to assess disease progression and survival for up to 12 months after the last dose of study drug. The total study duration will be dependent on overall patient tolerability to the study drug and response to treatment. It is anticipated that the duration of the entire study (Parts 1 and 2) could be approximately 3 years from first patient treated to last patient completed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, ages 12 years and older, with relapsed or refractory B-ALL who have failed, or are intolerant to, any established therapy; or for whom no other treatment options are available.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Serum/plasma creatinine ≤1.5mg/dL.
* Serum/plasma alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2 times the upper limit of normal (ULN); ≤5 times ULN if there is liver or bone involvement.
* Total serum/plasma bilirubin ≤1.5 times ULN.
* White Blood Cell Count value of <15,000 cells/μL prior to Cycle 1 Day 1.
* Negative urine or serum beta-human chorionic gonadotropin (β-HCG) pregnancy test within 7 days prior to the Cycle 1, Day 1 visit, for women of childbearing potential.
* Males, and female patients who are biologically capable of having children, must agree to use a medically acceptable method of birth control.

Exclusion Criteria:

* Patients who have an option for other treatment for B-ALL at the current state of disease.
* Known active central nervous system (CNS) leukemia.
* Patients with Burkitt's leukemia/lymphoma.
* Active graft-versus-host disease.
* Autologous or allogenic transplant within the 60 days prior to Screening.
* Known history of immunogenicity or hypersensitivity to a CD19 antibody.
* Known history of positive serum human ADA.
* Active autoimmune disease, motor neuropathy considered of autoimmune origin, or other central nervous system autoimmune disease.
* Known seropositive for human immunodeficiency (HIV) virus, hepatitis B surface antigen (HbsAg), or antibody to hepatitis C virus (anti-HCV).
* History of Stevens-Johnson syndrome or toxic epidermal necrolysis syndrome.
* Pregnant or breastfeeding women.
* Significant medical comorbidities, including uncontrolled hypertension (diastolic blood pressure >115 mm Hg), unstable angina, congestive heart failure (greater than New York Heart Association class II), severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia, poorly controlled diabetes, severe chronic pulmonary disease, coronary angioplasty, myocardial infarction within 6 months prior to Screening, or uncontrolled atrial or ventricular cardiac arrhythmias.
* Use of any other experimental medication(s) within 14 days or 5 half-lives, but in no case <14 days prior to the start of treatment on Cycle 1, Day 1, except if approved by the Sponsor.
* Major surgery, chemotherapy, systemic therapy (excluding hydroxyurea,steroids and any targeted small molecules or biologics), or radiotherapy, within 14 days or 5 half-lives (whichever is shorter) prior to the Cycle 1, Day 1 treatment, except if approved by the Sponsor.
* Failure to recover from acute non hematologic toxicity (except alopecia or Grade 2 or lower neuropathy), due to previous therapy, prior to Screening.
* Isolated extramedullary relapse.
* Congenital long QT syndrome or a corrected QTc interval of ≥450 ms at the Screening visit.
* Active second primary malignancy other than non-melanoma skin cancers, nonmetastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy determined not be exclusionary.
* Any other significant medical illness, abnormality, or condition that would make the patient inappropriate for study participation or put the patient at risk.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-03; Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Emory University Hospital, Atlanta, Georgia
  - The University of Chicago Medical Center, Chicago, Illinois
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University Hospital of Cleveland, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, James Cancer Hospital, Columbus, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jain N, Stock W, Zeidan A, Atallah E, McCloskey J, Heffner L, Tomlinson B, Bhatnagar B, Feingold J, Ungar D, Chao G, Zhang X, Qin Y, Havenith K, Kantarjian H, Wieduwilt MJ. Loncastuximab tesirine, an anti-CD19 antibody-drug conjugate, in relapsed/refractory B-cell acute lymphoblastic leukemia. Blood Adv. 2020 Feb 11;4(3):449-457. doi: 10.1182/bloodadvances.2019000767. PMID 32012214

RESULTS

PARTICIPANT FLOW:
Groups:
- 15 μg/kg Q3W: Participants received 15 μg/kg ADCT-402 on Day 1 of each 3-week treatment cycle.
- 30 μg/kg Q3W: Participants received 30 μg/kg ADCT-402 on Day 1 of each 3-week treatment cycle.
- 60 μg/kg Q3W: Participants received 60 μg/kg ADCT-402 on Day 1 of each 3-week treatment cycle.
- 90 μg/kg Q3W: Participants received 90 μg/kg ADCT-402 on Day 1 of each 3-week treatment cycle.
- 120 μg/kg Q3W: Participants received 120 μg/kg ADCT-402 on Day 1 of each 3-week treatment cycle.
- 150 μg/kg Q3W: Participants received 150 μg/kg ADCT-402 on Day 1 of each 3-week treatment cycle.
- 50 μg/kg QW: Participants received 50 μg/kg ADCT-402 weekly on Days 1, 8 and 15 of each 3-week (21-day) treatment cycle. This dose level for the weekly (QW) dosing schedule was based on the safety and tolerability of participants who had been treated on the every 3-week (Q3W) schedule.
Period: Overall Study
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W | 50 μg/kg QW
Started | 5 | 7 | 3 | 4 | 5 | 6 | 5
Completed | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not Completed | 5 | 6 | 3 | 3 | 5 | 6 | 5
Not completed — Death | 5 | 5 | 3 | 3 | 3 | 6 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Miscellaneous | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- 50 μg/kg QW: Participants received 50 μg/kg ADCT-402 on Days 1, 8 and 15 of each 3-week (21-day) treatment cycle. This dose level for the QW dosing was based on the safety and tolerability of participants who have been treated on the every 3-week (Q3W) schedule.
- Total: Total of all reporting groups
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W | 50 μg/kg QW | Total
Number analyzed (Participants) | 5 | 7 | 3 | 4 | 5 | 6 | 5 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (21.22) | 49.6 (21.95) | 50.3 (6.51) | 63.8 (7.09) | 46.8 (18.14) | 45.2 (19.61) | 42.8 (24.30) | 48.3 (18.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 1 | 2 | 4 | 4 | 16
  Male | 2 | 6 | 2 | 3 | 3 | 2 | 1 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 1 | 0 | 2 | 5 | 2 | 15
  Not Hispanic or Latino | 3 | 4 | 2 | 4 | 3 | 1 | 3 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 4 | 7 | 1 | 4 | 5 | 3 | 3 | 27
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 7 | 3 | 4 | 5 | 6 | 5 | 35
Height [Mean (Standard Deviation); unit: cm] — Population: Height data was not collected for 3 participants because of complications during the collection of baseline measurements.
  cm
    number analyzed (Participants) | 5 | 7 | 2 | 4 | 5 | 5 | 4 | 32
    (all) | 162.40 (8.510) | 167.97 (17.050) | 162.60 (0.000) | 164.78 (11.943) | 172.32 (10.146) | 163.58 (7.398) | 155.75 (5.072) | 164.83 (11.211)
Weight [Mean (Standard Deviation); unit: kg] | 76.44 (26.043) | 93.80 (31.551) | 87.13 (13.301) | 58.33 (15.745) | 78.00 (11.663) | 83.05 (38.842) | 70.58 (11.576) | 79.28 (25.631)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI could not be calculated for 3 participants due to missing height information.
  kg/m^2
    number analyzed (Participants) | 5 | 7 | 2 | 4 | 5 | 5 | 4 | 32
    (all) | 28.62 (7.192) | 34.05 (13.059) | 30.43 (3.504) | 21.07 (3.356) | 26.22 (2.949) | 32.70 (12.605) | 27.93 (5.741) | 29.15 (9.142)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Mean (Standard Deviation); unit: Score on a scale] — ECOG performance status is graded from 0 (fully active and able to carry on all pre-disease performance without restriction) to 5 (dead).
  Score on a scale | 1.00 (0.000) | 1.29 (0.488) | 0.67 (0.577) | 1.50 (0.577) | 1.60 (0.548) | 1.33 (1.033) | 1.40 (0.548) | 1.29 (0.622)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: A DLT is defined as any of the following events, except those that are clearly due to underlying disease or extraneous causes:
  A hematologic DLT is defined as:
  - Grade 3 or higher event of neutropenia or thrombocytopenia, or a Grade 4 anemia, with a hypocellular bone marrow lasting for 6 weeks or more after the start of a cycle, in the absence of residual leukemia (i.e., with <5% blasts). In case of a normocellular bone marrow with <5% blasts, 8 weeks with ≥Grade 3 pancytopenia will be considered a DLT.
  A non-hematologic DLT is defined as:
  * Grade 4 tumor lysis syndrome (Grade 3 TLS will not constitute DLT unless it leads to irreversible end-organ damage).
  * Grade 3 or higher AE (including nausea, vomiting, diarrhea, and electrolyte imbalances lasting more than 48 hours despite optimal therapy; excluding all grades of alopecia).
  * CTCAE Grade 3 or higher hypersensitivity reaction (regardless of premedication).
  * CTCAE Grade 3 or higher skin ulceration.
Time Frame: Day 1 to End of Cycle 1 (3 weeks)
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W | 50 μg/kg QW
Number analyzed (Participants) | 5 | 7 | 3 | 4 | 5 | 6 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0

2. Primary Outcome: Recommended Dose of ADCT-402 for Part 2
Description: The recommended dose was to be established by the dose escalation steering committee and based on safety findings during part 1 of the study.
Time Frame: Day 1 to End of Cycle 1 (3 weeks)
Population: This analysis was planned, but data was not collected as the study was terminated prematurely.
Groups:
- Part 1: ADCT-402 Dose Escalation: Weekly administration (QW) - Participants received an intravenous (IV) infusion of ADCT-402, on Days 1, 8, and 15 of each 3- week (21-day) cycle.
  3-week administration (Q3W) - Participants received an IV infusion of ADCT-402, on Day 1 of each 3-week (21-day) cycle.
  The dose escalation was conducted according to a 3+3 design.
Arm/Group | Part 1: ADCT-402 Dose Escalation
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Participants Reporting at Least One Treatment Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participants enrolled into this study regardless of its causal relationship to study drug. A TEAE is defined as any event not present before exposure to study drug or any event already present that worsens in either intensity or frequency after exposure to study drug.
Time Frame: From first dose of study drug up to 12 weeks after last dose (up to 39 weeks)
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W | 50 μg/kg QW
Number analyzed (Participants) | 5 | 7 | 3 | 4 | 5 | 6 | 5
Participants | 5 | 7 | 3 | 4 | 5 | 6 | 5

4. Primary Outcome: Number of Participants Reporting at Least One Treatment Emergent Serious Adverse Event (SAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant enrolled into this study regardless of its causal relationship to study drug. A treatment-emergent AE (TEAE) is defined as any event not present before exposure to study drug or any event already present that worsens in either intensity or frequency after exposure to study drug. An SAE is defined as any event that results in death, is immediately life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: From first dose of study drug up to 12 weeks after last dose (up to 39 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W | 50 μg/kg QW
Number analyzed (Participants) | 5 | 7 | 3 | 4 | 5 | 6 | 5
Participants | 5 | 4 | 2 | 3 | 5 | 5 | 4

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the number of participants with a best overall response of complete response (CR), complete response with incomplete blood count recovery (Cri) or partial response (PR) at the time each participant discontinues treatment with ADCT-402.
  CR is defined as achieving each of the following:
  * Bone marrow differential showing ≤5% blast cells.
  * Absolute neutrophil count (ANC) ≥1.0 x 10^9/L and platelet count ≥100 x 10^9/L.
  * Absence of extramedullary disease.
  * Participant is independent of red blood cell transfusions.
  Cri is defined as achieving all CR criteria except that values for ANC may be <1.0 x 10^9/L and/or values for platelets may be <100 x 10^9/L.
  PR is defined as achieving each of the following:
  * ANC ≥1.0 x 10^9/L and platelet count ≥100 x 10^9/L.
  * Bone marrow differential showing a ≥50% decrease from baseline in the percentage of bone marrow blast cells to a level >5% and ≤25%, or bone marrow differential showing <5% blast cells.
Time Frame: From 6 days prior to Day 1 of Cycle 3 and 5, and at each subsequent cycle, until discontinuation, assessed up to 12 months after last dose of study drug
Population: This analysis was planned, but data was not collected as the study was terminated prematurely.
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W | 50 μg/kg QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Duration of Response
Description: Duration of response is defined among responders (complete response [CR], complete response with incomplete blood count recovery [Cri], and partial response [PR]) as the time from the earliest date of first response until the first date of either disease progression or death due to any cause.
  Disease progression is defined as:
  * For participants with CR or CRi, the first date of reappearance of blast cells in bone marrow and/or peripheral blood to a level ≥5%, or development of extramedullary disease.
  * For participants with PR, the first date of an increase in blast cells in bone marrow and/or peripheral blood such that the patient does not continue to meet the criteria for PR.
Time Frame: as for outcome 5
Population: This analysis was planned, but data was not collected as the study was terminated prematurely.
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W | 50 μg/kg QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the first dose of study drug treatment until the date of death due to any cause.
Time Frame: as for outcome 5
Population: This analysis was planned, but data was not collected as the study was terminated prematurely.
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W | 50 μg/kg QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined among the efficacy population as the time from first dose of study drug until the first date of either disease progression or death due to any cause.
Time Frame: as for outcome 5
Population: This analysis was planned, but data was not collected as the study was terminated prematurely.
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W | 50 μg/kg QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for ADCT-402 Administered Every 3 Weeks (Q3W)
Description: Cmax for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the Q3W cohorts.
Time Frame: Day 1 (before infusion, end of infusion, and 1, 3 and 6 hours after infusion) and Days 2, 3, 5, 8 and 15 for Cycles 1 and 2
Population: Only participants with evaluable pharmacokinetic results were included in the analysis. Where data is not presented, the pharmacokinetic profiles were non-measurable or short-lived in duration; therefore, no analysis could be performed.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W
Number analyzed (Participants) | 5 | 7 | 3 | 4 | 5 | 6
µg/L
  PBD-Conjugated Ab : Cycle 1: number analyzed (Participants) | 4 | 7 | 3 | 3 | 5 | 6
  PBD-Conjugated Ab : Cycle 1 | 178 (128) | 258 (162) | 449 (282) | 1058 (893) | 1291 (1020) | 2145 (1054)
  PBD-Conjugated Ab : Cycle 2: number analyzed (Participants) | 1 | 4 | 2 | 2 | 5 | 4
  PBD-Conjugated Ab : Cycle 2 | 2150 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 339 (276) | 661 (412) | 1813 (1650) | 1515 (1001) | 3033 (1458)
  Total Ab (ADCT-402) : Cycle 1: number analyzed (Participants) | 4 | 7 | 2 | 3 | 4 | 6
  Total Ab (ADCT-402) : Cycle 1 | 205 (162) | 317 (194) | 717 (429) | 1049 (892) | 1722 (785) | 2761 (1718)
  Total Ab (ADCT-402) : Cycle 2: number analyzed (Participants) | 2 | 4 | 2 | 2 | 4 | 4
  Total Ab (ADCT-402) : Cycle 2 | 1251 (1724) | 366 (251) | 689 (382) | 1845 (1676) | 2125 (944) | 4338 (2460)
  SG3199 : Cycle 1: number analyzed (Participants) | 0 | 2 | 0 | 2 | 3 | 6
  SG3199 : Cycle 1 |  | 0.0428 (0.0000707) |  | 0.0617 (0.0238) | 0.0810 (0.0288) | 0.0907 (0.0500)
  SG3199 : Cycle 2: number analyzed (Participants) | 0 | 1 | 1 | 1 | 3 | 2
  SG3199 : Cycle 2 |  | 0.0459 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0697 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0551 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.108 (0.0239) | 0.0550 (0.0277)

10. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for ADCT-402 Administered Every Week (QW)
Description: Cmax for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the QW cohort.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | 50 μg/kg QW
Number analyzed (Participants) | 3
µg/L
  PBD-Conjugated Ab : Cycle 1 Week 1: number analyzed (Participants) | 1
  PBD-Conjugated Ab : Cycle 1 Week 1 | 777 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  PBD-Conjugated Ab : Cycle 1 Week 2: number analyzed (Participants) | 2
  PBD-Conjugated Ab : Cycle 1 Week 2 | 788 (456)
  PBD-Conjugated Ab : Cycle 1 Week 3: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 1: number analyzed (Participants) | 1
  PBD-Conjugated Ab : Cycle 2 Week 1 | 444 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  PBD-Conjugated Ab : Cycle 2 Week 2: number analyzed (Participants) | 1
  PBD-Conjugated Ab : Cycle 2 Week 2 | 757 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  PBD-Conjugated Ab : Cycle 2 Week 3: number analyzed (Participants) | 1
  PBD-Conjugated Ab : Cycle 2 Week 3 | 773 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab (ADCT-402): Cycle 1 Week 1 | 363 (390)
  Total Ab (ADCT-402): Cycle 1 Week 2 | 544 (492)
  Total Ab (ADCT-402): Cycle 1 Week 3: number analyzed (Participants) | 2
  Total Ab (ADCT-402): Cycle 1 Week 3 | 293 (313)
  Total Ab (ADCT-402): Cycle 2 Week 1: number analyzed (Participants) | 2
  Total Ab (ADCT-402): Cycle 2 Week 1 | 300 (294)
  Total Ab (ADCT-402): Cycle 2 Week 2: number analyzed (Participants) | 2
  Total Ab (ADCT-402): Cycle 2 Week 2 | 480 (414)
  Total Ab (ADCT-402): Cycle 2 Week 3: number analyzed (Participants) | 1
  Total Ab (ADCT-402): Cycle 2 Week 3 | 730 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  SG3199 : Cycle 1 Week 1: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 3: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 1: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 3: number analyzed (Participants) | 0

11. Secondary Outcome: Time to Reach the Maximum Serum Concentration (Tmax) for ADCT-402 Administered Every 3 Weeks (Q3W)
Description: Tmax for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the Q3W cohorts.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W
Number analyzed (Participants) | 4 | 7 | 3 | 3 | 5 | 6
days
  PBD-Conjugated Ab : Cycle 1 | 0.0525 (0.00957) | 0.0671 (0.0547) | 0.0433 (0.00577) | 0.0567 (0.0208) | 0.0460 (0.00548) | 0.0517 (0.00983)
  PBD-Conjugated Ab: Cycle 2: number analyzed (Participants) | 1 | 4 | 2 | 2 | 5 | 4
  PBD-Conjugated Ab: Cycle 2 | 0.0600 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0475 (0.0250) | 0.0300 (0.0141) | 0.0500 (0.0424) | 0.0500 (0.0212) | 0.0525 (0.0250)
  Total Ab (ADCT-402) : Cycle 1: number analyzed (Participants) | 4 | 7 | 2 | 3 | 4 | 6
  Total Ab (ADCT-402) : Cycle 1 | 0.0600 (0.0216) | 0.0729 (0.0547) | 0.0450 (0.00707) | 0.0433 (0.00577) | 0.0450 (0.00577) | 0.0517 (0.00983)
  Total Ab (ADCT-402) : Cycle 2: number analyzed (Participants) | 1 | 4 | 2 | 2 | 4 | 4
  Total Ab (ADCT-402) : Cycle 2 | 0.0600 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0700 (0.0678) | 0.0300 (0.0141) | 0.0500 (0.0424) | 0.0600 (0.0141) | 0.0625 (0.0263)
  SG3199 : Cycle 1: number analyzed (Participants) | 0 | 2 | 0 | 2 | 3 | 6
  SG3199 : Cycle 1 |  | 0.0600 (0.0283) |  | 0.125 (0.0636) | 0.0867 (0.00577) | 0.395 (0.777)
  SG3199 : Cycle 2: number analyzed (Participants) | 0 | 1 | 1 | 1 | 3 | 2
  SG3199 : Cycle 2 |  | 0.0600 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0600 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0400 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0867 (0.00577) | 0.0600 (0.0283)

12. Secondary Outcome: Time to Reach the Maximum Serum Concentration (Tmax) for ADCT-402 Administered Every Week (QW)
Description: Tmax for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the QW cohort.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 50 μg/kg QW
Number analyzed (Participants) | 3
days
  PBD-Conjugated Ab : Cycle 1 Week 1: number analyzed (Participants) | 1
  PBD-Conjugated Ab : Cycle 1 Week 1 | 0.0500 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  PBD-Conjugated Ab : Cycle 1 Week 2: number analyzed (Participants) | 2
  PBD-Conjugated Ab : Cycle 1 Week 2 | 0.0400 (0.0141)
  PBD-Conjugated Ab : Cycle 1 Week 3: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 1: number analyzed (Participants) | 1
  PBD-Conjugated Ab : Cycle 2 Week 1 | 0.0400 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  PBD-Conjugated Ab : Cycle 2 Week 2: number analyzed (Participants) | 1
  PBD-Conjugated Ab : Cycle 2 Week 2 | 0.0400 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  PBD-Conjugated Ab : Cycle 2 Week 3: number analyzed (Participants) | 1
  PBD-Conjugated Ab : Cycle 2 Week 3 | 0.0400 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab (ADCT-402): Cycle 1 Week 1 | 0.0500 (0.0100)
  Total Ab (ADCT-402): Cycle 1 Week 2 | 0.697 (1.14)
  Total Ab (ADCT-402): Cycle 1 Week 3: number analyzed (Participants) | 2
  Total Ab (ADCT-402): Cycle 1 Week 3 | 0.110 (0.0849)
  Total Ab (ADCT-402): Cycle 2 Week 1: number analyzed (Participants) | 2
  Total Ab (ADCT-402): Cycle 2 Week 1 | 0.0400 (0)
  Total Ab (ADCT-402): Cycle 2 Week 2: number analyzed (Participants) | 2
  Total Ab (ADCT-402): Cycle 2 Week 2 | 0.0300 (0.0141)
  Total Ab (ADCT-402): Cycle 2 Week 3: number analyzed (Participants) | 1
  Total Ab (ADCT-402): Cycle 2 Week 3 | 0.0400 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  SG3199 : Cycle 1 Week 1: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 3: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 1: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 3: number analyzed (Participants) | 0

13. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) for ADCT-402 Administered Every 3 Weeks (Q3W)
Description: AUClast for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the Q3W cohorts.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day*ug/L
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W
Number analyzed (Participants) | 4 | 7 | 3 | 3 | 5 | 6
day*ug/L
  PBD-Conjugated Ab : Cycle 1 | 337 (651) | 127 (229) | 43.0 (37.3) | 671 (1083) | 3907 (8159) | 688 (570)
  PBD-Conjugated Ab : Cycle 2: number analyzed (Participants) | 1 | 4 | 2 | 2 | 5 | 4
  PBD-Conjugated Ab : Cycle 2 | 1596 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 735 (1400) | 50.6 (9.08) | 3370 (4562) | 8744 (17745) | 7553 (727)
  Total Ab (ADCT-402) : Cycle 1: number analyzed (Participants) | 4 | 7 | 2 | 3 | 4 | 6
  Total Ab (ADCT-402) : Cycle 1 | 610 (1190) | 408 (623) | 59.9 (43.5) | 558 (899) | 5718 (9648) | 1091 (673)
  Total Ab (ADCT-402) : Cycle 2: number analyzed (Participants) | 2 | 4 | 2 | 2 | 4 | 4
  Total Ab (ADCT-402) : Cycle 2 | 1012 (1301) | 1140 (2096) | 40.2 (0.0244) | 3671 (5062) | 13519 (22799) | 10493 (2021)
  SG3199 : Cycle 1: number analyzed (Participants) | 0 | 2 | 0 | 2 | 3 | 6
  SG3199 : Cycle 1 |  | 0.00355 (0.00147) |  | 0.00930 (0.00675) | 0.0194 (0.0231) | 0.0338 (0.0150)
  SG3199 : Cycle 2: number analyzed (Participants) | 0 | 1 | 1 | 1 | 3 | 2
  SG3199 : Cycle 2 |  | 0.00522 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0129 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.00830 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.0433 (0.0316) | 0.00927 (0.00881)

14. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) for ADCT-402 Administered Every Week (QW)
Description: AUClast for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the QW cohort.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day*ug/L
Arm/Group | 50 μg/kg QW
Number analyzed (Participants) | 3
day*ug/L
  PBD-Conjugated Ab : Cycle 1 Week 1: number analyzed (Participants) | 1
  PBD-Conjugated Ab : Cycle 1 Week 1 | 518 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  PBD-Conjugated Ab : Cycle 1 Week 2: number analyzed (Participants) | 2
  PBD-Conjugated Ab : Cycle 1 Week 2 | 1063 (1334)
  PBD-Conjugated Ab : Cycle 1 Week 3: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 1: number analyzed (Participants) | 1
  PBD-Conjugated Ab : Cycle 2 Week 1 | 1548 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  PBD-Conjugated Ab : Cycle 2 Week 2: number analyzed (Participants) | 1
  PBD-Conjugated Ab : Cycle 2 Week 2 | 2631 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  PBD-Conjugated Ab : Cycle 2 Week 3: number analyzed (Participants) | 1
  PBD-Conjugated Ab : Cycle 2 Week 3 | 3918 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab (ADCT-402): Cycle 1 Week 1 | 464 (290)
  Total Ab (ADCT-402): Cycle 1 Week 2 | 821 (886)
  Total Ab (ADCT-402): Cycle 1 Week 3: number analyzed (Participants) | 2
  Total Ab (ADCT-402): Cycle 1 Week 3 | 1286 (1158)
  Total Ab (ADCT-402): Cycle 2 Week 1: number analyzed (Participants) | 2
  Total Ab (ADCT-402): Cycle 2 Week 1 | 1157 (962)
  Total Ab (ADCT-402): Cycle 2 Week 2: number analyzed (Participants) | 2
  Total Ab (ADCT-402): Cycle 2 Week 2 | 9.08 (9.78)
  Total Ab (ADCT-402): Cycle 2 Week 3: number analyzed (Participants) | 1
  Total Ab (ADCT-402): Cycle 2 Week 3 | 3927 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  SG3199 : Cycle 1 Week 1: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 3: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 1: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 3: number analyzed (Participants) | 0

15. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to Infinity (AUC∞) for ADCT-402 Administered Every 3 Weeks (Q3W)
Description: AUC∞ for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the Q3W cohorts.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day*ug/L
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W
Number analyzed (Participants) | 1 | 2 | 1 | 3 | 2 | 5
day*ug/L
  PBD-Conjugated Ab : Cycle 1: number analyzed (Participants) | 1 | 2 | 0 | 3 | 2 | 5
  PBD-Conjugated Ab : Cycle 1 | 1378 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 395 (371) |  | 677 (1091) | 282 (324) | 486 (259)
  PBD-Conjugated Ab : Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Total Ab (ADCT-402) : Cycle 1: number analyzed (Participants) | 0 | 2 | 1 | 1 | 0 | 2
  Total Ab (ADCT-402) : Cycle 1 |  | 535 (668) | 94.1 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 1634 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |  | 1140 (1283)
  Total Ab (ADCT-402) : Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  SG3199 : Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  SG3199 : Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to Infinity (AUC∞) for ADCT-402 Administered Weekly (QW)
Description: AUC∞ for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the QW cohort.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day*ug/L
Arm/Group | 50 μg/kg QW
Number analyzed (Participants) | 1
day*ug/L
  PBD-Conjugated Ab : Cycle 1 Week 1 | 545 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  PBD-Conjugated Ab : Cycle 1 Week 2: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 1 Week 3: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 1: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 2: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 3: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 1 Week 1: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 1 Week 2: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 1 Week 3: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 2 Week 1: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 2 Week 2: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 2 Week 3: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 1: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 3: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 1: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 3: number analyzed (Participants) | 0

17. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to the End of the Dosing Interval (AUC0-tau) for ADCT-402 Administered Every 3 Weeks (Q3W)
Description: AUCtau for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the Q3W cohorts.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day*ug/L
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W
Number analyzed (Participants) | 1 | 3 | 2 | 2 | 4 | 4
day*ug/L
  PBD-Conjugated Ab : Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  PBD-Conjugated Ab : Cycle 2 | 1810 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 985 (1606) | 53.3 (9.99) | 3595 (4876) | 8282 (14386) | 7444 (831)
  Total Ab (ADCT-402) : Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Total Ab (ADCT-402) : Cycle 2: number analyzed (Participants) | 1 | 3 | 1 | 1 | 4 | 4
  Total Ab (ADCT-402) : Cycle 2 | 2500 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 1607 (2330) | 41.2 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 7820 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 10198 (15433) | 10112 (1753)
  SG3199 : Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  SG3199 : Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  SG3199 : Cycle 2 |  |  |  |  | 0.104 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |

18. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to the End of the Dosing Interval (AUC0-tau) for ADCT-402 Administered Every Week (QW)
Description: AUCtau for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the QW cohort.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: day*ug/L
Arm/Group | 50 μg/kg QW
Number analyzed (Participants) | 2
day*ug/L
  PBD-Conjugated Ab : Cycle 1 Week 1: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 1 Week 2 | 1293 (1640)
  PBD-Conjugated Ab : Cycle 1 Week 3: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 1: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 2: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 3: number analyzed (Participants) | 1
  PBD-Conjugated Ab : Cycle 2 Week 3 | 3542 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab (ADCT-402): Cycle 1 Week 1: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 1 Week 2 | 1402 (1314)
  Total Ab (ADCT-402): Cycle 1 Week 3: number analyzed (Participants) | 1
  Total Ab (ADCT-402): Cycle 1 Week 3 | 2066 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab (ADCT-402): Cycle 2 Week 1: number analyzed (Participants) | 1
  Total Ab (ADCT-402): Cycle 2 Week 1 | 449 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab (ADCT-402): Cycle 2 Week 2: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 2 Week 3: number analyzed (Participants) | 1
  Total Ab (ADCT-402): Cycle 2 Week 3 | 3463 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  SG3199 : Cycle 1 Week 1: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 3: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 1: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 3: number analyzed (Participants) | 0

19. Secondary Outcome: Accumulation Index (AI) for ADCT-402 Administered Every 3 Weeks (Q3W)
Description: AI for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the Q3W cohorts. AI is the ratio of AUC 0-24 after multiple doses versus a single dose. It is the increase in drug plasma concentration after multiple dosing until a steady state is reached.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W
Number analyzed (Participants) | 1 | 3 | 1 | 1 | 3 | 4
ratio
  PBD-Conjugated Ab : Cycle 2 | 1.01 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 1.14 (0.242) | 1.00 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 1.06 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 1.30 (0.509) | 1.03 (0.0187)
  Total Ab (ADCT-402) : Cycle 2: number analyzed (Participants) | 1 | 2 | 1 | 1 | 2 | 3
  Total Ab (ADCT-402) : Cycle 2 | 1.04 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 1.62 (0.433) | 1.00 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 1.08 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 1.67 (0.939) | 1.06 (0.0532)
  SG3199 : Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Accumulation Index (AI) for ADCT-402 Administered Weekly (QW)
Description: AI for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the QW cohort. AI is the ratio of AUC 0-24 after multiple doses versus a single dose. It is the increase in drug plasma concentration after multiple dosing until a steady state is reached.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 50 μg/kg QW
Number analyzed (Participants) | 2
ratio
  PBD-Conjugated Ab : Cycle 1 Week 2 | 1.13 (0.0410)
  PBD-Conjugated Ab : Cycle 1 Week 3: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 2: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 3: number analyzed (Participants) | 0
  Total Ab (ADCT-402) : Cycle 1 Week 2 | 2.52 (1.92)
  Total Ab (ADCT-402) : Cycle 1 Week 3: number analyzed (Participants) | 0
  Total Ab (ADCT-402) : Cycle 2 Week 2: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 2 Week 3: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 3: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 3: number analyzed (Participants) | 0

21. Secondary Outcome: Volume of Distribution at Steady State for ADCT-402
Time Frame: as for outcome 9
Population: This analysis was planned, but data was not collected as the study was terminated prematurely.
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W | 50 μg/kg QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Mean Residence Time for ADCT-402
Time Frame: as for outcome 9
Population: This analysis was planned, but data was not collected as the study was terminated prematurely.
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W | 50 μg/kg QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Terminal Elimination Phase Rate Constant for ADCT-402
Time Frame: as for outcome 9
Population: This analysis was planned, but data was not collected as the study was terminated prematurely.
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W | 50 μg/kg QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Apparent Terminal Phase Elimination Half-life (T1/2) for ADCT-402 Administered Every 3 Weeks (Q3W)
Description: T1/2 for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the Q3W cohorts.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W
Number analyzed (Participants) | 1 | 3 | 1 | 3 | 3 | 5
days
  PBD-Conjugated Ab : Cycle 1: number analyzed (Participants) | 1 | 2 | 0 | 3 | 2 | 5
  PBD-Conjugated Ab : Cycle 1 | 5.23 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 1.87 (0.287) |  | 0.355 (0.501) | 0.156 (0.164) | 0.713 (0.596)
  PBD-Conjugated Ab : Cycle 2: number analyzed (Participants) | 1 | 3 | 1 | 1 | 3 | 4
  PBD-Conjugated Ab : Cycle 2 | 2.91 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 4.31 (6.62) | 0.282 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 4.96 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 7.55 (10.3) | 3.99 (0.723)
  Total Ab (ADCT-402) : Cycle 1: number analyzed (Participants) | 0 | 2 | 1 | 1 | 0 | 2
  Total Ab (ADCT-402) : Cycle 1 |  | 1.28 (1.66) | 0.0538 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.784 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |  | 0.275 (0.306)
  Total Ab (ADCT-402) : Cycle 2: number analyzed (Participants) | 1 | 2 | 1 | 1 | 2 | 3
  Total Ab (ADCT-402) : Cycle 2 | 4.42 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 15.0 (6.88) | 0.0342 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 5.59 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 14.5 (16.4) | 4.67 (1.68)
  SG3199 : Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  SG3199 : Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  SG3199 : Cycle 2 |  |  |  |  | 0.508 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |

25. Secondary Outcome: Apparent Terminal Phase Elimination Half-life (T1/2) for ADCT-402 Administered Every Week (QW)
Description: T1/2 for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the QW cohort.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 50 μg/kg QW
Number analyzed (Participants) | 2
days
  PBD-Conjugated Ab : Cycle 1 Week 1: number analyzed (Participants) | 1
  PBD-Conjugated Ab : Cycle 1 Week 1 | 2.29 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  PBD-Conjugated Ab : Cycle 1 Week 2 | 2.26 (0.288)
  PBD-Conjugated Ab : Cycle 1 Week 3: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 1: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 2: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 3: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 1 Week 1: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 1 Week 2 | 9.39 (9.77)
  Total Ab (ADCT-402): Cycle 1 Week 3: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 2 Week 1: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 2 Week 2: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 2 Week 3: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 1: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 3: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 1: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 3: number analyzed (Participants) | 0

26. Secondary Outcome: Apparent Clearance at Steady State for ADCT-402 Administered Every 3 Weeks (Q3W)
Description: Apparent clearance for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the Q3W cohorts.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: L/day
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 4 | 5
L/day
  PBD-Conjugated Ab : Cycle 1: number analyzed (Participants) | 1 | 2 | 0 | 3 | 2 | 5
  PBD-Conjugated Ab : Cycle 1 | 0.650 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 14.0 (14.3) |  | 80.8 (106) | 84.3 (102) | 27.4 (12.4)
  PBD-Conjugated Ab : Cycle 2: number analyzed (Participants) | 1 | 3 | 2 | 2 | 4 | 4
  PBD-Conjugated Ab : Cycle 2 | 0.495 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 69.3 (92.3) | 86.4 (34.6) | 9.63 (12.5) | 31.1 (37.0) | 1.57 (0.726)
  Total Ab (ADCT-402) : Cycle 1: number analyzed (Participants) | 0 | 2 | 1 | 1 | 0 | 2
  Total Ab (ADCT-402) : Cycle 1 |  | 31.3 (40.0) | 55.5 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 3.98 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |  | 18.9 (21.8)
  Total Ab (ADCT-402) : Cycle 2: number analyzed (Participants) | 1 | 3 | 1 | 1 | 4 | 4
  Total Ab (ADCT-402) : Cycle 2 | 0.422 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 16.4 (19.9) | 146 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 0.831 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 10.3 (16.7) | 1.37 (0.656)
  SG3199 : Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  SG3199 : Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  SG3199 : Cycle 2 |  |  |  |  | 838 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |

27. Secondary Outcome: Apparent Clearance at Steady State for ADCT-402 Administered Every Week (QW)
Description: Apparent clearance for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the QW cohort.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: L/day
Arm/Group | 50 μg/kg QW
Number analyzed (Participants) | 2
L/day
  PBD-Conjugated Ab : Cycle 1 Week 1: number analyzed (Participants) | 1
  PBD-Conjugated Ab : Cycle 1 Week 1 | 5.77 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  PBD-Conjugated Ab : Cycle 1 Week 2 | 14.0 (18.0)
  PBD-Conjugated Ab : Cycle 1 Week 3: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 1: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 2: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 3: number analyzed (Participants) | 1
  PBD-Conjugated Ab : Cycle 2 Week 3 | 1.01 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab (ADCT-402): Cycle 1 Week 1: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 1 Week 2 | 5.23 (5.16)
  Total Ab (ADCT-402): Cycle 1 Week 3: number analyzed (Participants) | 1
  Total Ab (ADCT-402): Cycle 1 Week 3 | 2.03 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab (ADCT-402): Cycle 2 Week 1: number analyzed (Participants) | 1
  Total Ab (ADCT-402): Cycle 2 Week 1 | 8.46 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  Total Ab (ADCT-402): Cycle 2 Week 2: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 2 Week 3: number analyzed (Participants) | 1
  Total Ab (ADCT-402): Cycle 2 Week 3 | 1.21 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  SG3199 : Cycle 1 Week 1: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 3: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 1: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 3: number analyzed (Participants) | 0

28. Secondary Outcome: Apparent Volume of Distribution (Vd Beta) for ADCT-402 Administered Every 3 Weeks (Q3W)
Description: Vd beta for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the Q3W cohorts.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W
Number analyzed (Participants) | 1 | 3 | 1 | 3 | 3 | 5
liters
  PBD-Conjugated Ab : Cycle 1: number analyzed (Participants) | 1 | 2 | 0 | 3 | 2 | 5
  PBD-Conjugated Ab : Cycle 1 | 4.91 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 40.7 (44.3) |  | 10.5 (12.6) | 6.89 (3.13) | 34.2 (35.5)
  PBD-Conjugated Ab : Cycle 2: number analyzed (Participants) | 1 | 3 | 1 | 1 | 3 | 4
  PBD-Conjugated Ab : Cycle 2 | 2.08 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 24.0 (18.1) | 45.1 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 5.61 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 8.33 (5.43) | 9.45 (5.27)
  Total Ab (ADCT-402) : Cycle 1: number analyzed (Participants) | 0 | 2 | 1 | 1 | 0 | 2
  Total Ab (ADCT-402) : Cycle 1 |  | 9.77 (1.09) | 4.31 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 4.50 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |  | 2.68 (0.309)
  Total Ab (ADCT-402) : Cycle 2: number analyzed (Participants) | 1 | 2 | 1 | 1 | 2 | 3
  Total Ab (ADCT-402) : Cycle 2 | 2.69 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 145 (190) | 7.22 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 6.71 (NA) — Standard deviation could not be determined as only one participant had evaluable data. | 11.4 (0.101) | 9.14 (5.96)
  SG3199 : Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  SG3199 : Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  SG3199 : Cycle 2 |  |  |  |  | 614 (NA) — Standard deviation could not be determined as only one participant had evaluable data. |

29. Secondary Outcome: Apparent Volume of Distribution (Vd Beta) for ADCT-402 Administered Every Week (QW)
Description: Vd beta for Pyrrolobenzodiazepine (PBD) conjugated antibody (Ab), total Ab and free warhead (SG3199) for the QW cohort.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | 50 μg/kg QW
Number analyzed (Participants) | 2
liters
  PBD-Conjugated Ab : Cycle 1 Week 1: number analyzed (Participants) | 1
  PBD-Conjugated Ab : Cycle 1 Week 1 | 19.1 (NA) — Standard deviation could not be determined as only one participant had evaluable data.
  PBD-Conjugated Ab : Cycle 1 Week 2 | 49.5 (64.6)
  PBD-Conjugated Ab : Cycle 1 Week 3: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 1: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 2: number analyzed (Participants) | 0
  PBD-Conjugated Ab : Cycle 2 Week 3: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 1 Week 1: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 1 Week 2 | 107 (144)
  Total Ab (ADCT-402): Cycle 1 Week 3: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 2 Week 1: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 2 Week 2: number analyzed (Participants) | 0
  Total Ab (ADCT-402): Cycle 2 Week 3: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 1: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 1 Week 3: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 1: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 2: number analyzed (Participants) | 0
  SG3199 : Cycle 2 Week 3: number analyzed (Participants) | 0

30. Secondary Outcome: Number of Participants With Anti-drug Antibody Response (ADA) Against ADCT-402
Description: Blood serum samples were collected and analysed to determine the presence or absence of ADA.
Time Frame: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: ADCT-402 Dose Escalation
Number analyzed (Participants) | 35
Participants
  Confirmed positive ADA pre-dose | 1
  Confirmed positive ADA post-dose | 0
  Confirmed positive ADA at any time | 1

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 12 weeks after last dose (up to 39 weeks)
Arm/Group | 15 μg/kg Q3W | 30 μg/kg Q3W | 60 μg/kg Q3W | 90 μg/kg Q3W | 120 μg/kg Q3W | 150 μg/kg Q3W | 50 μg/kg QW
All-Cause Mortality (participants affected / at risk) | 5/5 | 5/7 | 3/3 | 3/4 | 3/5 | 6/6 | 3/5
Serious Adverse Events (participants affected / at risk) | 5/5 | 4/7 | 2/3 | 3/4 | 5/5 | 5/6 | 4/5
Other Adverse Events (participants affected / at risk) | 5/5 | 7/7 | 3/3 | 4/4 | 5/5 | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 15 μg/kg Q3W (N=5) | 30 μg/kg Q3W (N=7) | 60 μg/kg Q3W (N=3) | 90 μg/kg Q3W (N=4) | 120 μg/kg Q3W (N=5) | 150 μg/kg Q3W (N=6) | 50 μg/kg QW (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 2 | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Candida sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungaemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blast cells present (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 15 μg/kg Q3W (N=5) | 30 μg/kg Q3W (N=7) | 60 μg/kg Q3W (N=3) | 90 μg/kg Q3W (N=4) | 120 μg/kg Q3W (N=5) | 150 μg/kg Q3W (N=6) | 50 μg/kg QW (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 1 | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 3 | 5 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 3 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angina bullosa haemorrhagica (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 3 | 1 | 3 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 3 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 2 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 2 | 2 | 4 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 2 | 3 | 3 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 2 | 2 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 1 | 1 | 3 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 2 | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 2 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 2 | 0 | 0 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 1
White blood cell count decreased (Investigations) | 0 | 2 | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Amylase decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspergillus test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
High density lipoprotein decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 1 | 0 | 2 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 2 | 2 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 2 | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 3
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was early terminated prior to part 2 because of slow accrual. Formal assessment of potential anti-leukemic effect was not undertaken because of the early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can publish after first multi-site publication, or if no multi-site publication is made within 18 months of study completion/termination. The only disclosure restriction on the PI is the sponsor can review results comms. prior to public release and can embargo comms. regarding trial results for a period that is more than 60 but less than or equal to 180 days from the time submitted to sponsor for review. The sponsor can't require changes to the communication and can't extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT02669264/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT02669264/SAP_001.pdf